CLINICAL TRIAL: NCT01360047
Title: Association Between Low Dose Acetylsalicylic Acid (ASA) and Proton Pump Inhibitors and Risk of Acute Myocardial Infarction or Coronary Heart Disease Death - Nested Case Control Analyses in a Cohort of First-time Users of Low Dose ASA for Secondary Prevention of Cerebrovascular and Cardiovascular Outcomes.
Brief Title: Association Between Low Dose Acetylsalicylic Acid (ASA) and Proton Pump Inhibitors and Risk of Acute Myocardial Infarction or Coronary Death
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D961FN00006
Record Dates: First submitted 2011-05-24; First posted 2011-05-25 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Nonfatal Myocardial Infarction; Coronary Death
Keywords: MI; low dose aspirin; PPI; epidemiology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Cases: Cases with nonfatal MI or coronary death
- Controls: Age, sex, and calendar-year matched controls sampled from the original study cohort to be a round number of at least four times the number of cases

SUMMARY:
The purpose of this study is to estimate the risk of myocardial infarction (MI)/coronary death associated with use of monotherapy low dose ASA (single antiplatelet) as well as concomitant use of monotherapy low dose ASA and proton pump inhibitors (PPIs) in first- time users of low dose ASA for secondary prevention using a UK primary care database.

DETAILED DESCRIPTION:
Number of Anticipated Subjects: In case-control analysis 5.000-10.000

ELIGIBILITY:
Inclusion Criteria:

* As above (study population description).
* All individuals aged 50-84 years with at least two year of enrolment with the primary care physician (PCP) and a computerized prescription history of at least one year before the start of the study.

Exclusion Criteria:

* Recorded diagnosis of cancer prior to study start.
* Alcohol abuse or alcohol-related disease prior to study start.
* Patients aged ≥ 70 years with a follow-up longer than one year if having fewer than two recorded consultations with a primary care physician (PCP) during their entire follow-up (proxy for incomplete and invalid data recording) which for some individuals will be close to 8 years.

Ages: 50 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients aged 50 to 84 years with a first ever prescription of low-dose ASA (defined as 75-300 mg/day) for the secondary prevention of cardiovascular or cerebrovascular events (defined as any previous ischemic cerebrovascular event or ischemic heart disease) from 1 January 2000 to 31 December 2007.
Sampling Method: Non-Probability Sample
Enrollment: 39513 (Actual)
Dates: Start 2011-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Nonfatal MI or coronary death | Up to eight years from entry into study cohort

CONTACTS AND LOCATIONS:
Overall Officials: Luis A Garcia Rodriguez, Principal Investigator — CEIFE (Centro Español de Investigación Farmacoepidemiológica)
Locations (1):
- Research Site, Madrid, Spain